CLINICAL TRIAL: NCT05459935
Title: Treatment of Pediatric Hypertrophic Tonsils and Pediatric Obstructive Sleep Apnea by Non-invasive Photobiomodulation
Brief Title: Photobiomodulation for Pediatric Hypertrophic Tonsils
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00103330
Record Dates: First submitted 2022-05-19; First posted 2022-07-15 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Pediatric Sleep Apnea; Obstructive Sleep Apnea; Tonsils Hypertrophy
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant
Masking Description: Sham intervention (nonactivated/unpowered phototherapy intervention)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- PBM Tonsil Arm (Experimental): Photobiomodulation exposure of hypertrophic tonsils
  Interventions: Device: PBM Tonsil Arm
- Tonsil Control Arm (Sham Comparator): Sham (non-powered) exposure of hypertrophic tonsils
  Interventions: Device: Sham PBM Tonsil Arm

INTERVENTIONS:
Device: PBM Tonsil Arm — exposure of hypertrophic tonsils to photobiomodulation
  Other Names: Fotona Lightwalker AT S
  Arms: PBM Tonsil Arm
Device: Sham PBM Tonsil Arm — non-powered exposure of hypertrophic tonsils to photobiomodulation
  Other Names: Fotona Lightwalker AT S - non-powered
  Arms: Tonsil Control Arm

SUMMARY:
Pediatric obstructive sleep apnea is a medical condition where a child has great difficulty with breathing, or stops breathing all together, while asleep. This is a medical condition for which the primary treatment is usually a surgery targeted towards removing swollen tonsils and adenoids. However, surgical removal of tonsils and adenoids comes with its own risks of complications during and after surgery including secondary hemorrhage and long term increased risks for respiratory and infectious diseases. Perhaps more importantly, surgical removal of swollen tonsils and adenoids does not guarantee successful treatment of a child's obstructive sleep apnea.

The use of laser light therapy in a non-cutting manner (known as photobiomodulation and abbreviated as PBM) has been a relatively new development within medicine. Recently, dentists have begun to use PBM as a method to treat adult snoring and, with lesser success, adult obstructive sleep apnea. To date, there are no known side effects to the use of PBM for the treatment of any sleep breathing disorders. However, no research has been published on the use of PBM for the treatment of pediatric obstructive sleep apnea or swollen tonsils in children

The purpose of this project is to determine whether photobiomodulation can provide a beneficial effect on pediatric hypertrophic tonsils and pediatric obstructive sleep apnea and, if it does, to create the appropriate workflow, referral pathways, and treatment parameters for clinicians to provide this treatment as a multidisciplinary approach in a clinical setting.

The investigators hypothesize that photobiomodulation can be used successfully to decrease the pediatric hypertrophic tonsils in children with symptoms of an pediatric obstructive sleep apnea and will also result in improved AHI scores (be able to breath significantly better when sleeping) in these children.

ELIGIBILITY:
Inclusion Criteria:

* Brodsky visually graded tonsils 3/4
* patient must assent, parent must consent, to all pre and post follow up including sleep testing
* patient and parent must agree to normal referral protocols regardless of participation within this study or not

Exclusion Criteria:

* visual indication of cancerous growth
* currently under treatment (pharmacologic, other) for hypertrophic tonsils
* already scheduled for surgical intervention of hypertrophic tonsils

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 64 (Estimated)
Dates: Start 2022-10-15 (Actual); Primary Completion 2026-07-06 (Estimated); Study Completion 2030-01-06 (Estimated)

PRIMARY OUTCOMES:
Tonsil Size | immediately after intervention
  Tonsil size grading (Brodsky score): 0-4, 0 being not present 4 being restrictive to entire airway. Lower scores are better. Each integer represents 25% obstruction of airway (0 being not visible, 1 being 0-25%, 2 being 25-50%, 3 being 50-75%, 4 being 75-100%). There is no abbreviated scale title.

SECONDARY OUTCOMES:
AHI Score | Next Day (next night)
  Comparisons of before and after AHI score by portable sleep testing device
Questionnaire Improvement | night after, per quarter after for 1 year
  Comparisons of before and after PSQ (pediatric sleep questionnaire) scores

CONTACTS AND LOCATIONS:
Locations (1):
- Enjoy Dental, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No